CLINICAL TRIAL: NCT05144165
Title: Systemic Treatment of Moderate-to-severe Psoriasis in Adults: Update of the French Guidelines Using Delphi Consensus Statement
Brief Title: Systemic Treatment of Moderate-to-severe Psoriasis in Adults: Update of the French Guidelines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre of Evidence of the French Society of Dermatology (Other)
Responsible Party: Sponsor
Other Study IDs: CDPDelphiPso
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Psoriasis; Psoriasis Palmaris; Psoriasis Inverse; Psoriasis Vulgaris; Psoriatic Nail; Psoriatic Plaque; Psoriasis Guttate; Psoriasis of Scalp; Psoriasis Universalis; Psoriatic Erythroderma; Psoriasis Pustular
Keywords: Delphi; Consensus statement; Guidelines; Experts
MeSH Terms: conditions — Psoriasis; Guttate Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Experts consensus — Consensus opinion using Delphi Methodology

SUMMARY:
French guidelines on the use of systemic treatments for moderate-to-severe psoriasis in adults have been developed by the psoriasis research group of the French Society of Dermatology using literature available until July 2017 (Amatore et al, 2019). Because several systemic treatments have been marketed since then, new guidelines are mandatory. The aim of this study coordinated by the Centre of Evidence of the French Society of Dermatology is to update the available French guidelines using a Delphi method.

DETAILED DESCRIPTION:
Justification of Delphi methodology

The Delphi method has been widely used for elaboration of guidelines. The goal of the Delphi method is to solicit group opinion and to combine the opinion of a panel of experts into a consensus (or dissensus). During a Delphi study, multiple rounds of questionnaires are sent to a panel of experts with feedback between rounds, allowing experts to re-evaluate their responses along with the replies of other experts.

Design, expert eligibility and data collection A steering committee of members of the French Centre of Evidence (G. Chaby, F. Corgibet, L. Fardet, S. Leducq, F. Poizeau https://reco.sfdermato.org/fr/centre-de-preuves-en-dermatologie) and members of the Psoriasis Research Group of the French Society of Dermatology (M. Chastagner, L. Gouillon), without any competing interest regarding this topic, will be in charge with elaboration and conduction of the Delphi study.

The selected experts will be asked whether they agree to participate in the Delphi survey. Upon acceptance, they will be asked to answer the Delphi study administered using the online survey Welphi®. Before the first round, demographic information (age, sex, location of practice, availability of a phototherapy cabin, public or private practice) and competing interests will be collected. All experts will provide informed consent. Experts will have 2 weeks to complete the online survey with two email reminders. For each round, the number of experts who completed the surveys will be documented.

Procedure

Definition of consensus For statements with responses on an ordinal 7-point Likert scale (rating 1, strongly disagree to 7 strongly agree), 'agreement' will be defined as a score of 5-7, 'neutral' by a score of 4 and 'disagreement' by a score of 1-3. Consensus will be defined as achieved when > 70% experts will vote for a given option on the Likert scale. For Multiple Choice Questions (MCQs), consensus will be defined as achieved if > 70% experts voted for a particular option. Median and interquartile range (IQR) will be used to describe the central tendency and dispersion of responses: a "strong statement" will be defined as a median score of ≥ 6 or ≤ 2 on the Likert scale and 90% votes for MCQs. If consensus is not reached for one question (using Likert scale or MCQ) after 3 rounds, dissensus is acted. For this study, four rounds are planned, including round 1 with open-ended questions (see below) and a maximum of three rounds to obtain consensus.

ELIGIBILITY:
Inclusion criteria

* French dermatologists
* public and private practice practitioners
* members of the French Society of Dermatology
* expertise in the field of psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the Centre of Evidence (M. Beylot-Barry, G. Chaby, O. Chosidow, F. Corgibet, L. Fardet, B. Guillot, N. Jouan, D. Jullien) will propose a list of 40 to 50 French dermatologists experts in the field of psoriasis. Members of the scientific committees of the psoriasis research group (French Society of Dermatology) and "Resopso" will be included in the list of experts, with the exception of those participating of the design and publication of the present study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Update of the French guidelines by consensus using participating experts opinions | 15 days to complete the online survey for each round
  Round 1 will include
  * 3 questions using an ordinal 7-point Likert scale, regarding every systemic treatment that could be prescribed as a first, second or subsequent line, in patients with moderate-to-severe plaque psoriasis without contra-indication to any treatment
  * 9 questions using an ordinal 7-point Likert scale, regarding first line therapeutic management of particular forms of psoriasis
  * 11 open-ended questions for special indications of each therapeutic agent.
  Round 2, 3 and 4 Experts will be asked to review the questionnaire based on the information provided in the former round. They will have to re-rate the 12 questions using the 7-point Likert scales. Regarding special indications for each therapeutic agent, expert's comments from round 1 will be synthesized and converted into MCQs for subsequent rounds. If consensus is reached for one question, the question will not reappear in subsequent rounds.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Evidence of Dermatology, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Amatore F, Villani AP, Tauber M, Viguier M, Guillot B; Psoriasis Research Group of the French Society of Dermatology (Groupe de Recherche sur le Psoriasis de la Societe Francaise de Dermatologie). French guidelines on the use of systemic treatments for moderate-to-severe psoriasis in adults. J Eur Acad Dermatol Venereol. 2019 Mar;33(3):464-483. doi: 10.1111/jdv.15340. Epub 2019 Feb 22. PMID 30793796
- See also: French Centre of Evidence in Dermatology — https://centredepreuves.sfdermato.org